CLINICAL TRIAL: NCT03409965
Title: Evaluation of the Lutronic Infini and Lutronic LaseMD Systems in Combination Treatment
Brief Title: Lutronic Infini and LaseMD Systems in Combination Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L17002
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Face and Neck Wrinkles, Texture, Pigmentation
MeSH Terms: conditions — Facies

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lutronic Systems Combination Treatment (Experimental): Combination treatment of the face and/or neck using the Lutronic Infini System and Lutronic LaseMD System.
  Interventions: Device: Lutronic Infini System; Device: Lutronic LaseMD System

INTERVENTIONS:
Device: Lutronic Infini System — A microneedle radiofrequency device
Device: Lutronic LaseMD System — A fractional thulium laser device

SUMMARY:
This is a prospective, multi-site, non-randomized study evaluating the safety and effectiveness of the Infini and LaseMD Systems for combination treatment in wrinkles, texture, and pigmentation of the face and/or neck.

DETAILED DESCRIPTION:
Enrolled subjects will receive three (3) face and/or neck treatments provided 30 days apart. During each treatment subjects will receive both Infini and LaseMD treatments. Treatments will be provided according to a protocol-specific treatment protocol in which an Infini treatment will be provided first, followed by a LaseMD treatment. A telephone contact will be completed at 3 days following each treatment to assess for adverse events. One follow-up visit will be conducted at 90 days following the last study treatment. Outcome measures include clinician grading and subject satisfaction post-treatment. Pre-treatment study photographs and D90 study photographs will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years and older.
2. Subject in good health.
3. Fitzpatrick Skin Type I to VI.
4. Solar elastosis on the face and/or neck.
5. Mild to moderate wrinkles of the face and/or neck.
6. Mild to moderate textural concerns on the face and/or neck.
7. Sun and/or age-related pigmentation on the face and/or neck.
8. Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
9. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
10. Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

    1. Postmenopausal for at least 12 months prior to study;
    2. Without a uterus and/or both ovaries; or
    3. Bilateral tubal ligation at least six months prior to study enrollment.
11. Absence of physical or psychological conditions unacceptable to the investigator.
12. Willingness to refrain from use of aspirin, Ibuprofen, Naproxen, or any other NSAID prior to each study treatment and chronic use during the entire post-treatment study period. Washout period, if chronic user, for 4 weeks prior to the first treatment. After all study treatments are completed, limited acute NSAID use is allowed, i.e., a maximum of 2-3 doses in any 2-week period, if needed.
13. Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
14. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Presence of an active systemic or local skin disease that may affect wound healing.
2. History of keloids or poor wound healing.
3. Severe solar elastosis.
4. Excessive subcutaneous fat in the area(s) to be treated.
5. Excessive skin laxity on the area(s) to be treated.
6. Significant scarring in the area(s) to be treated that would interfere with assessing results.
7. Open wounds or lesions in the area(s) to be treated.
8. Inability to understand the protocol or to give informed consent.
9. Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within four weeks prior to study participation or during the study.
10. Excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
11. BMI equal to or greater than 30.
12. History of chronic drug or alcohol abuse.
13. History of collagen vascular disease.
14. History of autoimmune disease.
15. Subjects with implanted pacemaker or defibrillator.
16. Subjects with sensitivity or allergy to gold.
17. Subjects with sensitivity or allergy to pre-treatment medication.
18. Subjects with photosensitive skin.
19. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
20. Subjects who anticipate the need for inpatient surgery or overnight hospitalization during the study.
21. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
22. Concurrent enrollment in any study involving the use of investigational devices or drugs.
23. Current smoker or history of smoking in the last five years.
24. Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
25. History of surgical or cosmetic treatments in the area(s) to be treated within the past year.
26. History or current use of the following prescription medications:

    1. Accutane or other systemic retinoids within the past twelve months;
    2. Topical Retinoids within the past two weeks; and/or
    3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix) within the past two weeks.
27. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Masked, qualitative assessment of improvement | 90 days following the last study treatment
  An assessment of paired pre- and post-treatment photographs will be conducted by blinded assessors. Each blinded assessor will be given an identical set of baseline (pre-treatment) and Day 90 follow-up photos to be assessed. Each photo's visit interval, i.e., pre-treatment and follow-up, will NOT be marked. Each blinded assessor will conduct their assessment independently, comparing the Left and Right photos for improvement in the face and/or neck using the following definition:
  * Change: An improvement that is:
  * Striking, substantial and immediately noticeable, or
  * Readily apparent but modest in nature
  * Slight and subtle in nature, may require close examination
  The assessor chooses the photo they believe to be the post-treatment photo, i.e., Left photo or Right photo.

SECONDARY OUTCOMES:
Clinician assessment of overall aesthetic improvement | 90 days following the last treatment.
  Overall aesthetic improvement based on completion of the Clinician Global Aesthetic Improvement Scale, a scale that rates global aesthetic improvement from the pretreatment appearance using the following definitions:
  1. = Improved: Improvement in appearance from initial condition
  2. = No Change: The appearance is essentially the same as the original condition
  3. = Worse: The appearance is worse than the original condition The scale will be administered based on a live assessment of the subject while referring to the subject's pre-treatment photographs, and based on a comparison of the subject's pre-treatment photographs to the Day 90 follow-up photographs.
Subject assessment of overall aesthetic improvement | 90 days following the last treatment.
  Overall aesthetic improvement based on completion of the Subject Global Aesthetic Improvement Scale, a scale that rates global aesthetic improvement from the pretreatment appearance using the following definitions:
  1. = Improved: Improvement in appearance from initial condition
  2. = No Change: The appearance is essentially the same as the original condition
  3. = Worse: The appearance is worse than the original condition Subjects will complete the scale based on a live assessment while referring to a hand mirror and their pre-treatment photographs, and based on a comparison of their pre-treatment photographs to their Day 90 follow-up photographs.
Patient Satisfaction | 90 days following study treatment
  Patient satisfaction will be evaluated based on subjects' completion of a patient satisfaction questionnaire while referring to a hand mirror and their pre-treatment photographs and their Day 90 follow-up photographs. Subjects will be asked to document Yes/No as to whether they notice any improvement in how their treated skin areas look; specify any changes they see in the treated areas, e.g., skin texture improvement, skin tone improvement, skin pigmentation improvement, etc.; characterize their level of satisfaction with study treatment based on 5 levels of satisfaction: Very satisfied, Satisfied, Slightly Satisfied, Neither Satisfied or Dissatisfied, Dissatisfied; document Yes/No if they would recommend the treatment to friends and family members.
Treatment-related pain | For the duration of each study treatment
  During study treatments, subjects' pain levels will be monitored using a validated Numeric Rating Scale (0-10), with 0 being 'No Pain' and 10 being the 'Worst Possible Pain'.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Larson, MBA, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - Moradi M.D., Vista, California
  - The Aesthetic Clinique, Santa Rosa Beach, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moradi A, Weiner SF. Effectiveness of Combining High-Intensity Focused Radiofrequency and Non-Ablative Fractional Laser for Improving the Appearance of the Aging Face and Neck. J Drugs Dermatol. 2019 Jan 1;18(1):59-64. PMID 30681798